CLINICAL TRIAL: NCT04096625
Title: Enhancement of a Psychotherapeutic Intervention Through Transcranial Direct Current Stimulation (tDCS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Stephan T. Egger, Senior Psychiatrists, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS ATP
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Psychiatric Disorder
Keywords: Brain Stimulation, tDCS, Psychotherapy, Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: The investigators plan a double-blind, randomised, sham-controlled trial in a cross-over design to assess the efficacy and safety of tDCS as an add-on intervention to a psychotherapeutic treatment for patients with a severe psychiatric condition requiring hospitalization.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS (Experimental): Active tDCS will be delivered at 2mA for 20 minutes.
  Interventions: Device: Active tDCS; Behavioral: Assertiveness Training Program (ATP); Device: Sham tDCS
- Sham tDCS (Sham Comparator): Sham tDCS: after 40 seconds of stimulation (2mA), a small current pulse was delivered every 550 msec (110 muA over 15 msec).
  Interventions: Device: Active tDCS; Behavioral: Assertiveness Training Program (ATP); Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS will be delivered at 2mA for 20 minutes.
Behavioral: Assertiveness Training Program (ATP) — The Assertiveness Training Program (ATP) is a cognitive-behavioural therapy delivered in group sessions.
Device: Sham tDCS — Sham tDCS, after 40 seconds of stimulation (2mA), a small current pulse was delivered every 550 msec (110 muA over 15 msec).

SUMMARY:
Transcranial Direct Current Stimulation (tDCS), is a neuromodulatory technique, that is safe, well-tolerated, easy to administer and fairly inexpensive. Results from tDCS trials involving participants with several neuropsychiatric disorders, including major depression, bipolar disorder, schizophrenia and substance use disorder are encouraging. The clinical effects of tDCS are broad; the underlying condition, the areas stimulated together with the type and duration of stimulation are important factors. In patients with neuropsychiatric conditions, a reduction of symptoms, an enhancement of neurocognitive functions together with an overall improvement in functionality and wellbeing have been consistently reported. These effects emerge during the stimulation period, in the weeks after stimulation, the effects seem to peak and consolidate further. tDCS appears to enhance the effects of other interventions as well; however, to date, there have been no studies into the effects of using tDCS as an add-on intervention to psychotherapy on symptoms and wellbeing

ELIGIBILITY:
Inclusion Criteria:

* Participants are competent to give informed consent, as determined by the referring physician or psychiatrist.
* German language proficiency as a native speaker or level B1
* A psychiatric diagnosis according to ICD-10;
* Three or more psychiatric hospitalizations in the past 12 months; or
* A cumulative length of stay over 40 days; or
* Referral for further treatment to our treatment unit.

Exclusion Criteria:

* Concomitant group psychotherapeutic intervention.
* Current neurological disorder.
* Current cardiovascular disorder.
* Current respiratory disorder.
* Current substance use or withdrawal.
* Epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychopathological Assessment | Change: Baseline, 3, 6 weeks, 6 and 12 months
  Symptom Questionnaire

SECONDARY OUTCOMES:
Insecurity- Self-confidence | Change: Baseline, 3, 6 weeks, 6 and 12 months
  Symptom Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stephan T. Egger, MD, Principal Investigator — Psychiatric University Hospital of Zurich
Locations (1):
- Psychiatrische Universitätsklinik Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No